CLINICAL TRIAL: NCT06427187
Title: Outcomes of Mechanical Thrombectomy of Acute Ischemic Stroke Anterior Circulation Distal Vessel Occlusion
Brief Title: Mechanical Thrombectomy of Acute Ischemic Stroke Anterior Circulation Distal Vessel Occlusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Zayed Saber, assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mechanical throbectomy
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Each presenting Patient subjected to:
  * careful history including Age, Sex, comorbid diseases (hypertension, Diabetes, dyslipidemia, cardiac disease...), time from onset to treatment
  * examination: Vital signs
  * NIHSS at admission
  * Lab investigation: basic lab, metabolic profile & Lipid profile
  * The diagnosis was made using a standard CT stroke protocol including CT head Aspect score, arterial CT angiography, and perfusion CT. In some cases, primary stroke MRI was performed including fluid attenuated inversion recovery (FLAIR), diffusion weighted imaging (DWI): in order to evaluate location of occluded vessel, size of ischemic core & penumbra).
  All patients received either mechanical thrombectomy (MT) with or without intra-venous thrombolysis (IVT) according to standard medical guidelines. MT was performed using approved aspiration catheters or stent-retrievers or both.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- distal vessel occlusion Mechanical thromectomy (Experimental): Each presenting Patient with acute distal vessel occlusion of anterior circulation with (A1-A3)or (M2-M3) either mechanical thrombectomy (MT) with or without intra-venous thrombolysis (IVT) according to standard medical guidelines. MT was performed using approved aspiration catheters or stent-retrievers or both.
  Interventions: Device: an array of devices are used in thrombectomy. These include guide catheters, stent-retrievers, microcatheters, aspiration catheters, and aspiration pump systems

INTERVENTIONS:
Device: an array of devices are used in thrombectomy. These include guide catheters, stent-retrievers, microcatheters, aspiration catheters, and aspiration pump systems — each patient with distal vessel occlusion subjected to mechanical thrombectomy using aspiration technique or stent retriever

SUMMARY:
Ischemic stroke continues to be of the leading causes of disability and death. Distal vessel occlusion one of most presenting and disabling varieties of ischemic stroke. Distal vessel occlusion stroke is a type of ischemic stroke that affects the small arteries in the brain, usually beyond the M2 segment of the middle cerebral artery. These strokes can cause various neurological symptoms depending on the location and size of the occluded vessel and the extent of the brain tissue damage

DETAILED DESCRIPTION:
DMVOs are defined by the Distal Thrombectomy Summit Group consensus statement as thromboembolic occlusion of the anterior cerebral artery, M2-M4 middle cerebral artery (MCA), posterior cerebral artery (PCA), posterior inferior cerebellar artery, anterior inferior cerebellar artery or superior cerebellar artery. It is estimated that 25-40% of all AIS is due to DMVO.Though distal vessel occlusion associated with poor disabling comorbidities'.With different aetiology weather primary Embolic from (heart, carotid or aorta),thrombotic (atherosclerotic, hypertension or Diabetes ,smoking &hyperlipidaemia) or Secondary distal vessel occlusion that occurs as a complication of a proximal large vessel occlusion, either spontaneously or after treatment with intravenous thrombolysis or endovascular thrombectomy. This can be due to thrombus fragmentation and migration or incomplete reperfusion of the affected vascular territory . Endovascular thrombectomy is well established as a highly effective treatment for acute ischemic stroke (AIS) due to proximal, large vessel occlusions (PLVOs). Recent advances in stent retriever and aspiration catheter technology are more promising results to reach more distal vessels, with a good outcome. However, MT in M2 emerging with different technique using stent Retriever or aspiration or both nowadays, evidence of other MT in distal vessel occlusion is poor.

ELIGIBILITY:
Inclusion Criteria:

* a. Inclusion criteria:

  1. Diagnosis of an acute ischemic stroke due to an occlusion of the anterior cerebral artery (ACA) in the A1-A3 segment 2. Diagnosis of an acute ischemic stroke due to an occlusion of the middle cerebral artery in the distal M2 segment or the M3 segment.

Exclusion Criteria:

1. Posterior circulation small vessel occlusion
2. Tandem lesions with occlusion of the ipsilateral ICA were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Thrombolysis in Cerebral Infarction (TICI) | 1 day , 10 day
  The original description was based on the angiographic appearances of the treated occluded vessel and the distal branches:
  grade 0: no perfusion grade 1: penetration with minimal perfusion grade 2: partial perfusion grade 2A: only partial filling (less than two-thirds) of the entire vascular territory is visualized grade 2B: complete filling of all of the expected vascular territory is visualized but the filling is slower than normal grade 3: complete perfusion
modified Thrombolysis in Cerebral Infarction scale (mTICI) | 1 day , 10 day
  grade 0: no perfusion grade 1: antegrade reperfusion past the initial occlusion, but limited distal branch filling with little or slow distal reperfusion grade 2 grade 2a: antegrade reperfusion of less than half of the occluded target artery previously ischemic territory (e.g. in one major division of the middle cerebral artery (MCA) and its territory) grade 2b: antegrade reperfusion of more than half of the previously occluded target artery ischemic territory (e.g. in two major divisions of the MCA and their territories) grade 2c: near complete perfusion except for slow flow or distal emboli in a few distal cortical vessels this was not part of the original mTICI score, but was added later and has since become widely accepted as being part of the scoring 4 grade 3: complete antegrade reperfusion of the previously occluded target artery ischemic territory, with absence of visualized occlusion in all distal branches

SECONDARY OUTCOMES:
mRS | three months
  90 Days modified Rankin scale (mRS) score The Modified Rankin Scale (mRS) is used to measure the degree of disability in patients who have had a stroke, as follows 0: No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Safety outcomes were defined as 90-day mortality and occurrence of symptomatic intracranial haemorrhage (sICH). | three months
  Safety outcomes were defined as 90-day mortality and occurrence of symptomatic intracranial haemorrhage (sICH).

REFERENCES:
- [Background] Kunz WG, Almekhlafi MA, Goyal M. Distal Vessel Occlusions: When to Consider Endovascular Thrombectomy. Stroke. 2018 Jul;49(7):1581-1583. doi: 10.1161/STROKEAHA.118.021887. Epub 2018 Jun 18. No abstract available. PMID 29915118
- [Background] Sepp D, Hernandez Petzsche MR, Zarth T, Wunderlich S, Ikenberg B, Maegerlein C, Zimmer C, Berndt MT, Boeckh-Behrens T, Kirschke JS. Mechanical thrombectomy of distal cerebral vessel occlusions of the anterior circulation. Sci Rep. 2023 Apr 7;13(1):5730. doi: 10.1038/s41598-023-32634-0. PMID 37029202
- [Background] Saver JL, Chapot R, Agid R, Hassan A, Jadhav AP, Liebeskind DS, Lobotesis K, Meila D, Meyer L, Raphaeli G, Gupta R; Distal Thrombectomy Summit Group*dagger. Thrombectomy for Distal, Medium Vessel Occlusions: A Consensus Statement on Present Knowledge and Promising Directions. Stroke. 2020 Sep;51(9):2872-2884. doi: 10.1161/STROKEAHA.120.028956. Epub 2020 Aug 6. No abstract available. PMID 32757757
- [Background] Kobeissi H, Bilgin C, Ghozy S, Kadirvel R, Kallmes DF, Brinjikji W. A review of acute ischemic stroke caused by distal, medium vessel occlusions. Interv Neuroradiol. 2025 Dec;31(6):846-851. doi: 10.1177/15910199231197616. Epub 2023 Aug 29. PMID 37644821
- [Background] Lima FO, Furie KL, Silva GS, Lev MH, Camargo EC, Singhal AB, Harris GJ, Halpern EF, Koroshetz WJ, Smith WS, Nogueira RG. Prognosis of untreated strokes due to anterior circulation proximal intracranial arterial occlusions detected by use of computed tomography angiography. JAMA Neurol. 2014 Feb;71(2):151-7. doi: 10.1001/jamaneurol.2013.5007. PMID 24323077
- [Background] Elhorany M, Rosso C, Shotar E, Baronnet-Chauvet F, Premat K, Lenck S, Crozier S, Corcy C, Bottin L, Mansour OY, Talbi A, El-Din EAT, Fadel WA, Sourour NA, Alamowitch S, Samson Y, Clarencon F. Safety and effectiveness of mechanical thrombectomy for primary isolated distal vessel occlusions: A monocentric retrospective comparative study. J Neuroradiol. 2022 Jun;49(4):311-316. doi: 10.1016/j.neurad.2022.03.008. Epub 2022 Apr 6. PMID 35397949
- [Background] Guenego A, Mine B, Bonnet T, Elens S, Vazquez Suarez J, Jodaitis L, Ligot N, Naeije G, Lubicz B. Thrombectomy for distal medium vessel occlusion with a new generation of Stentretriever (Tigertriever 13). Interv Neuroradiol. 2022 Aug;28(4):444-454. doi: 10.1177/15910199211039926. Epub 2021 Sep 13. PMID 34516332
- [Background] Alawieh AM, Chalhoub RM, Al Kasab S, Jabbour P, Psychogios MN, Starke RM, Arthur AS, Fargen KM, De Leacy R, Kan P, Dumont TM, Rai A, Crosa RJ, Maier I, Goyal N, Wolfe SQ, Cawley CM, Mocco J, Tjoumakaris SI, Howard BM, Dimisko L, Saad H, Ogilvy CS, Crowley RW, Mascitelli JR, Fragata I, Levitt MR, Kim JT, Park MS, Gory B, Polifka AJ, Matouk C, Grossberg JA, Spiotta AM; STAR Collaborators. Multicenter investigation of technical and clinical outcomes after thrombectomy for distal vessel occlusion by frontline technique. J Neurointerv Surg. 2023 Sep;15(e1):e93-e101. doi: 10.1136/jnis-2022-019023. Epub 2022 Aug 2. PMID 35918129
- [Background] Sweid A, Head J, Tjoumakaris S, Xu V, Shivashankar K, Alexander TD, Dougherty JA, Gooch MR, Herial N, Hasan D, DePrince M, Rosenwasser RH, Jabbour P. Mechanical Thrombectomy in Distal Vessels: Revascularization Rates, Complications, and Functional Outcome. World Neurosurg. 2019 Oct;130:e1098-e1104. doi: 10.1016/j.wneu.2019.07.098. Epub 2019 Jul 16. PMID 31323418
- [Background] Atchaneeyasakul K, Malik AM, Yavagal DR, Haussen DC, Jadhav AP, Bouslama M, Kenmuir CL, Desai S, Grossberg JA, Chaturvedi S, Jovin TG, Nogueira RG. Thrombectomy Outcomes in Acute Ischemic Stroke due to Middle Cerebral Artery M2 Occlusion with Stent Retriever versus Aspiration: A Multicenter Experience. Interv Neurol. 2020 Jan;8(2-6):180-186. doi: 10.1159/000500198. Epub 2019 Jun 18. PMID 32508900
- [Background] Sacks D, Baxter B, Campbell BCV, Carpenter JS, Cognard C, Dippel D, Eesa M, Fischer U, Hausegger K, Hirsch JA, Hussain MS, Jansen O, Jayaraman MV, Khalessi AA, Kluck BW, Lavine S, Meyers PM, Ramee S, Rufenacht DA, Schirmer CM, Vorwerk D. Multisociety Consensus Quality Improvement Revised Consensus Statement for Endovascular Therapy of Acute Ischemic Stroke: From the American Association of Neurological Surgeons (AANS), American Society of Neuroradiology (ASNR), Cardiovascular and Interventional Radiology Society of Europe (CIRSE), Canadian Interventional Radiology Association (CIRA), Congress of Neurological Surgeons (CNS), European Society of Minimally Invasive Neurological Therapy (ESMINT), European Society of Neuroradiology (ESNR), European Stroke Organization (ESO), Society for Cardiovascular Angiography and Interventions (SCAI), Society of Interventional Radiology (SIR), Society of NeuroInterventional Surgery (SNIS), and World Stroke Organization (WSO). J Vasc Interv Radiol. 2018 Apr;29(4):441-453. doi: 10.1016/j.jvir.2017.11.026. Epub 2018 Mar 1. No abstract available. PMID 29478797
- [Background] Zaidat OO, Yoo AJ, Khatri P, Tomsick TA, von Kummer R, Saver JL, Marks MP, Prabhakaran S, Kallmes DF, Fitzsimmons BF, Mocco J, Wardlaw JM, Barnwell SL, Jovin TG, Linfante I, Siddiqui AH, Alexander MJ, Hirsch JA, Wintermark M, Albers G, Woo HH, Heck DV, Lev M, Aviv R, Hacke W, Warach S, Broderick J, Derdeyn CP, Furlan A, Nogueira RG, Yavagal DR, Goyal M, Demchuk AM, Bendszus M, Liebeskind DS; Cerebral Angiographic Revascularization Grading (CARG) Collaborators; STIR Revascularization working group; STIR Thrombolysis in Cerebral Infarction (TICI) Task Force. Recommendations on angiographic revascularization grading standards for acute ischemic stroke: a consensus statement. Stroke. 2013 Sep;44(9):2650-63. doi: 10.1161/STROKEAHA.113.001972. Epub 2013 Aug 6. No abstract available. PMID 23920012